CLINICAL TRIAL: NCT04542668
Title: An Open-label, Randomized, Cross-over Study to Investigate the Effect of Weight-bearing vs Non-weight-bearing Exercise and Cardiovascular Stress Without Load on Collagen and Proteoglycan in Serum and Urine in Patients With Osteoarthritis
Brief Title: The Effect of Exercise on Serum Levels of Collagen and Proteoglycan in Patients With Knee Osteoarthritis
Acronym: EFEX-OA-02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordic Bioscience A/S (Industry)
Collaborators: University of Copenhagen (Other); NBCD A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: EFEX-OA-02_FINAL_Protocol_v1.2
Record Dates: First submitted 2020-08-27; First posted 2020-09-09 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The study period will be 4 weeks. In each week, the subjects will undergo a different physical activity intervention. The order of the interventions will be randomized. The interventions will be separated by a minimum of 4 days. Inteventions: Cycling, Running, exercise-simulation with inotropy and resting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cycling as first intervention (Other): Cycling -> Running -> Inotropy -> Resting
  Interventions: Other: Cycling then running; Other: Inotropy; Other: Resting
- Running as first intervention (Other): Running -> Cycling -> Inotropy -> Resting
  Interventions: Other: Running then cycling; Other: Inotropy; Other: Resting

INTERVENTIONS:
Other: Cycling then running — Ergometer cycling Treadmill running
  Other Names: Exercise
  Arms: Cycling as first intervention
Other: Running then cycling — Treadmill running Ergometer cycling
  Other Names: Exercise
  Arms: Running as first intervention
Other: Inotropy — Adrenaline induced inotropy
  Other Names: Exercise simulation
Other: Resting — Subjects must be minimally physically active
  Other Names: Non-Ex

SUMMARY:
The aim of EFEX-OA-02 is to explore how running, cycling, exercise simulation and resting acutely influence collagen and proteoglycan homeostasis in OA, as reflected by changes in collagen and proteoglycan levels in urine and serum.

ELIGIBILITY:
Inclusion Criteria:

1. Cumulated Osteoarthritis Kellgren-Lawrence radiological grade of at least 2 in the tibio-femoral joints diagnosed by screening X-ray.
2. 40 to < 75 years of age at time of signing the informed consent.
3. Body weight > 50 and < 100 kg and BMI in the range 18.5-35 kg/m2 .
4. Male or female.
5. Able to attend all four study sessions and comply with the dietary and activity restrictions.
6. Able to provide informed consent

Exclusion Criteria:

Medical conditions:

1. Osteoarthritis Kellgren-Lawrence radiological grade of 4 in one or both knees.
2. Cumulated osteoarthritis Kellgren-Lawrence radiological grade no higher than 1.
3. History of arthroscopy or intra-articular administration of corticosteroids or hyaluronic acid into the target knee within 6 months before screening.
4. Previous arthroplasty of knee or hip.
5. Intention to have major surgery during the timeframe of the study.
6. Secondary OA related to e.g. any known trauma including cruciate ligament tears, meniscus tears and cartilage damage, dysplasia, aseptic osteonecrosis, acromegaly, Paget disease, Stickler syndrome, hemochromatosis, gout, chondrocalcinosis (pseudogout).
7. Current treatment with beta-receptor adrenergic antagonists (beta-blockers), MAO inhibitor, systemic corticosteroid treatment in doses equivalent to > 10 mg prednisolone per day, or vitamin K antagonists, new oral anticoagulants, fractionated and non-fractionated heparin.
8. Active systemic infection.
9. Active systemic inflammatory or autoimmune disease.
10. Any sign of previous or current cardiovascular disease.
11. Not currently an active athlete or highly trained individual.

Other exclusion criteria:

1. Legal incapacity or limited legal capacity.
2. Inability to communicate or cooperate with the investigator or to comply with the requirements of the entire study.
3. Categorized as being very difficult to draw blood from, as evaluated by the investigator.
4. Current alcohol abuse and/or inability to refrain from intake of alcoholic beverages for 24 hours prior to the study intervention.
5. Other factors, e.g. self-reported drug abuse, which in the opinion of the investigator may interfere with the performance of the study.
6. Site staff, study staff members and study staff family members.
7. Other concomitant disease compromising or otherwise significantly affecting ECM turnover in the opinion of the investigator.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Acute chances in biomarkers | Acute: 0-4 hours and subacute: 24 hours
  Serum and urine biochemical markers of joint related collagens and proteoglycan (not further specified)

CONTACTS AND LOCATIONS:
Overall Officials: Niels Secher, MD, DMSci, Principal Investigator — University of Copenhagen
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No